CLINICAL TRIAL: NCT00771212
Title: Observational Study on the Patients With Pain Medications
Status: Completed | Type: Observational
Sponsor: Johnson & Johnson Taiwan Ltd (Industry)
Responsible Party: Sponsor
Other Study IDs: CR014656
Record Dates: First submitted 2008-10-10; First posted 2008-10-13 (Estimated); Last update posted 2014-05-23 (Estimated); Status verified 2014-05

CONDITIONS: Pain
Keywords: Pain; Observational; Taiwan
MeSH Terms: conditions — Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- 001
  Interventions: Other: Observational pain control study

INTERVENTIONS:
Other: Observational pain control study — Observational pain control study

SUMMARY:
The purpose of this study is to describe the use of pain treatments in Taiwan, the demographics, clinical characteristics of patients requiring pain treatments, current treatments, outcomes of treatments and the reasons for changing pain medication during treatment.

DETAILED DESCRIPTION:
This is a Phase IV, multi-center, observational study to describe the use of pain treatments, the demographics, clinical characteristics of patients requiring pain treatments, current treatments, outcomes of treatments and the reasons for changing pain medication during treatment. The study is conducted in an effort to understand the status of pain control in Taiwan. Currently in Taiwan, there is no approved documentation showing the most effective standard medication for treatment of patients in pain. Observational study with no study medication administered.

ELIGIBILITY:
Inclusion Criteria:

* Outpatients only
* Patients must have pain, previously treated with and without medication and have a VAS (Visual analogue scale) score recorded at the enrolment time
* Patient must have a VAS score >4

Exclusion Criteria:

* Patients who are receiving any investigational drug during the study
* Patients with known or suspected psychotic disease or mental retardation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Outpatients; Patients must have pain, previously treated with and without medication and have a VAS (Visual analogue scale) score recorded at the enrolment time; Patient must have a VAS score >4
Sampling Method: Probability Sample
Enrollment: 2636 (Actual)
Dates: Start 2007-10; Primary Completion 2008-05 (Actual); Study Completion 2008-05 (Actual)

PRIMARY OUTCOMES:
To describe effective use of pain medications, describe demographics, clinical characteristics of patients requiring pain treatments, current treatments, outcomes of treatments and the reasons for changing pain medication during treatment in Taiwan | 60 days

SECONDARY OUTCOMES:
Pain Relief Rating Scale | 60 days
Sleeping quality Assessment | 60 days
Global Assessments (Patient/Investigator) | 60 days

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Taiwan, Ltd. Clinical Trial, Study Director — Johnson & Johnson Taiwan Ltd